CLINICAL TRIAL: NCT00340600
Title: Continuation of Follow-up of DES-Exposed Cohorts
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998017; OH98-C-N017
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Autoimmune Disease; Prostate Cancer; Ovarian Cancer; Endometrial Cancer
Keywords: Cancer; DES; Endocrine Disrupting Chemicals; In Utero
MeSH Terms: conditions — Breast Neoplasms; Autoimmune Diseases; Prostatic Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- DES Exposed: DES-exposed mothers, daughters and sons, and identified subjects
- DES Unexposed: DES-unexposed mothers, daughters and sons, and identified subjects

SUMMARY:
Diethylstilbestrol (DES), a drug first synthesized in 1938, was administered to several million pregnant women in the U.S. and Europe for the prevention of spontaneous abortion and premature delivery. In 1971, Herbst reported a strong association between DES use in pregnancy and the occurrence of vaginal clear cell adenocarcinoma (CCA) in exposed female offspring. Animal models have demonstrated a range of DES effects on offspring exposed in utero, including reproductive dysfunction, immune system changes, behavioral and sexual abnormalities, and increases in various reproductive cancers in males and females. In the mid-1970's, several separate cohorts of DES-exposed daughters and unexposed comparison groups were followed for the occurrence of cancer, precursor lesions, and reproductive effects, but systematic follow-up of these cohorts had ceased by 1990. In 1992, Congress passed a bill (H;.R. 4178) mandating the continued follow-up of DES-exposed cohorts. The National Cancer Institute, in collaboration with five field centers, reassembled previously studied cohorts of DES-exposed and unexposed mothers, daughters and sons, and identified subjects with documented exposure status who had not been studied previously, through familial links within the cohorts. Standardized baseline questionnaires were mailed to cohort members to ascertain the risk of cancer and other disorders. Pathology reports were collected for reported cancers and preneoplastic conditions. Two separate rounds of follow up have been conducted and a third is almost complete. Patients from the Registry for Research on Hormonal Transplacental Carcinogenesis (the Registry) will be added to the follow-up effort in the third phase. The purpose of this study is to continue the follow-up, by means of mail questionnaires and medical record collection, which was begun during the first phase of the study. Concern has arisen that DES-exposed daughters may be at higher risk of breast cancer. Exposure to high levels of endogenous estrogen in utero has been hypothesized to increase the risk of breast cancer and DES is a potent estrogen. Cancer risk in the sons will also continue to be assessed, especially for increased risks of prostate cancer. Since the offspring who were exposed to DES in utero are currently reaching their late forties, when cancer rates begin to rise, it is important to continue the follow-up of these cohorts to determine if there are long-term increases in cancer risk.

DETAILED DESCRIPTION:
Diethylstilbestrol (DES), a drug first synthesized in 1938, was administered to several million pregnant women in the U.S. and Europe for the prevention of spontaneous abortion and premature delivery. In 1971, Herbst reported a strong association between DES use in pregnancy and the occurrence of vaginal clear cell adenocarcinoma (CCA) in exposed female offspring. Animal models have demonstrated a range of DES effects on offspring exposed in utero, including reproductive dysfunction, immune system changes, behavioral and sexual abnormalities, and increases in various reproductive cancers in males and females. In the mid-1970's, several separate cohorts of DES-exposed daughters and unexposed comparison groups were followed for the occurrence of cancer, precursor lesions, and reproductive effects, but systematic follow-up of these cohorts had ceased by 1990. In 1992, Congress passed a bill (H;.R. 4178) mandating the continued follow-up of DES-exposed cohorts of mothers, daughters, sons and grandchildren. The National Cancer Institute, in collaboration with five field centers, reassembled previously studied cohorts of DES-exposed and unexposed mothers, daughters and sons, and identified subjects with documented exposure status who had not been studied previously, through familial links within the cohorts. Standardized baseline questionnaires were mailed to cohort members to ascertain the risk of cancer and other disorders. Pathology reports were collected for reported cancers and preneoplastic conditions. Three separate phases of follow up have been conducted. Patients from the Registry for Research on Hormonal Transplacental Carcinogenesis at the University of Chicago will be added to the follow-up effort and mailed the questionaire used in the third phase of follow-up. A cohort of daughters of women exposed and not exposed to DES in utero have been added to the study to assess the effects of DES on third generation women.

The purpose of this study as a whole is to continue the follow-up, by means of mailed questionnaires and medical record collection, which was begun during the first phase of the study. Concern has arisen that DES-exposed daughters may be at higher risk of breast cancer. Exposure to high levels of endogenous estrogen in utero has been hypothesized to increase the risk of breast cancer and DES is a potent estrogen. Cancer risk in the sons will also continue to be assessed, especially for increased risks of prostate cancer. Since the offspring who were exposed to DES in utero are currently reaching their late forties, when cancer rates begin to rise, it is important to continue the follow-up of these cohorts to determine if there are long-term increases in cancer risk.

We are planning to add a biospecimen collection component to the study. We propose to conduct a pilot study, nested within our ongoing combined cohort of DES-daughters, at Boston University to determine the feasibility of recruiting women participating in our study for phlebotomy and to investigate potential differences in the hormone metabolites and methylation patterns of germline DNA in 60 of these samples representing three groups of women: those exposed to high doses of DES prenatally, those exposed to low-doses of DES prenatally, and unexposed. Hormone metabolites and DNA methylation will be assessed in relation to DES exposure. Hormone metabolites will be measured at NCI s Frederick laboratory. DNA methylation will be assessed by Dr. Shuk-Mei Ho, the Jacob G. Schmidlapp Chair of the Department of Environmental Health, Director of the Center for Environmental Genetics, and Co-Leader of the Hormonal Malignancies Program in the Joint Cancer Center, at the College of Medicine in the University of Cincinnati, OH, and at Stephen Chanock s laboratory at NCI. The findings of this pilot study may have profound implications for the mechanisms by which endocrine disruption in the fetus influences human health. IRB approval of the data collection protocol has been received from Boston University.

ELIGIBILITY:
* INCLUSION CRITERIA:

Exposed daughters and unexposed daughters originally identified at: Baylor College of Medicine, University of Southern California (USC), Gunderson Clinic, Mayo Clinic, and Massachusetts General Hospital (MGH).

Male and female offspring of mothers who were enrolled in a clinical trial to assess the effectiveness of DES at the University of Chicago.

Offspring of mothers who were treated with DES by an infertility specialist, Dr. Herbert Horne, in the Boston area.

Offspring of DES-exposed mothers and unexposed mothers who were followed for breast cancer risk during the 1980s.

Exposed sons and unexposed sons who were originally identified and followed at the Mayo Clinic during the late1970's for the occurrence of cancer, genital abnormalities and infertility.

Subjects from the Registry for Research on Hormonal Transplacental Carcinogenesis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DES-exposed and unexposed mothers, daughters and sons, and identified subjects
Sampling Method: Non-Probability Sample
Enrollment: 10805 (Actual)
Dates: Start 1998-03-18 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Cancer | With Each Follow-up
  primary outcome is cancer

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Troisi, D.Sc., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Boston University School of Public Health, Boston, Massachusetts, United States

REFERENCES:
- [Background] Robboy SJ, Noller KL, O'Brien P, Kaufman RH, Townsend D, Barnes AB, Gundersen J, Lawrence WD, Bergstrahl E, McGorray S, et al. Increased incidence of cervical and vaginal dysplasia in 3,980 diethylstilbestrol-exposed young women. Experience of the National Collaborative Diethylstilbestrol Adenosis Project. JAMA. 1984 Dec 7;252(21):2979-83. PMID 6502858
- [Background] Labarthe D, Adam E, Noller KL, O'Brien PC, Robboy SJ, Tilley BC, Townsend D, Barnes AB, Kaufman RH, Decker DG, Fish CR, Herbst AL, Gundersen J, Kurland LT. Design and preliminary observations of National Cooperative Diethylstilbestrol Adenosis (DESAD) Project. Obstet Gynecol. 1978 Apr;51(4):453-8. doi: 10.1097/00006250-197804000-00014. PMID 662228
- [Background] Herbst AL, Ulfelder H, Poskanzer DC. Adenocarcinoma of the vagina. Association of maternal stilbestrol therapy with tumor appearance in young women. N Engl J Med. 1971 Apr 22;284(15):878-81. doi: 10.1056/NEJM197104222841604. No abstract available. PMID 5549830